CLINICAL TRIAL: NCT05266469
Title: Exploring the Characteristics and Profiles of Relapsing Multiple Sclerosis Patients Initiated on Ofatumumab or Ocrelizumab in a Real-World Setting in the Gulf Region
Brief Title: Exploring the Profiles of RMS Patients on Ofatumumab or Ocrelizumab in a Real-World Setting in the Gulf
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GAE01
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; RMS; NIS; Gulf Region; Ofatumumab; Ocrelizumab
MeSH Terms: interventions — ofatumumab; ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ofatumumab: Patients prescribed with Ofatumumab
  Interventions: Other: Ofatumumab
- Ocrelizumab: Patients prescribed with Ocrelizumab
  Interventions: Other: Ocrelizumab

INTERVENTIONS:
Other: Ofatumumab — There is no treatment allocation. Patients administered Ofatumumab by prescription will be enrolled.
  Groups: Ofatumumab
Other: Ocrelizumab — There is no treatment allocation. Patients administered Ocrelizumab by prescription will be enrolled.
  Groups: Ocrelizumab

SUMMARY:
This is a retrospective and prospective, observational mixed-methods (quantitative and qualitative) cohort study of patients who are treated with either Ofatumumab or Ocrelizumab that will be recruited and followed up for one year to collect their profiles across the Gulf countries.

DETAILED DESCRIPTION:
This study will be conducted retrospectively (for patients who had their first treatment initiated on either Ofatumumab or Ocrelizumab before study start and from 2019 onwards) and prospectively (for patients who are initiated on either drug during the active recruitment period which spans for one year after the start of the first data collection) using data collected in a standardized manner.

Index date (baseline): Defined as the date of the first treatment initiated on either Ofatumumab or Ocrelizumab Index period: The patients fulfilling the inclusion criteria will be identified during the recruitment period (01-Jan-2019 to 01-April-2023 or up to 1 year after the start of the active recruitment period).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females.
* Age 18 to 65 years.
* Confirmed RMS diagnosis as per the 2017 updated McDonald's criteria (Thompson et al., 2018).
* Having their first dose of either drugs during the index period (2019 onwards and up to 1 year since start of the active recruitment period).
* The decision to initiate either drug should be based on the patient's disease and taken by the treating physician before the decision of inviting the patient to participate in the study.
* The patient agreed and provided informed consent on the use of his/her de-identified data.

Exclusion Criteria:

* Patients below 18 years or above 65 years.
* Pregnant females.
* SPMS and/or PPMS patients.
* The patient's refusal to be included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males and Females aged 18 to 65 years with a confirmed RMS diagnosis, and a provided agreement on the shared informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Baseline
  EDSS: Score 0 to 10, with 0 as "Normal Neurological Exam" and 10 as "Death Due to MS
Magnetic Resonance Imaging (MRI) activity | Baseline
  number of participants with:
  * T1-Gd+
  * absence of T1-Gd+
  * T2 lesions
Volume of T2 lesions | Baseline
  Volume of T2 lesions will be provided
Number of relapses in the past 12 months | Baseline
  Number of relapses in the past 12 months will be collected. Relapse is defined as the occurrence of new symptoms or the worsening of old symptoms that happens during the Multiple Sclerosis course
Baseline ARR (Annualized Relapse Rates) | Baseline
  Baseline ARR (Annualized Relapse Rates) will be collected
Time since MS diagnosis | Baseline
  Time since Multiple Sclerosis (MS) diagnosis will be provided
Time since first MS symptom | Baseline
  Time since first Multiple Sclerosis (MS) symptom will be collected
Percentage of participants with previous DMTs | Baseline
  Percentage of participants with previous Disease modifying therapies (DMTs) will be collected
Time from diagnosis to start of treatment | Baseline
  Time from diagnosis to start of treatment will be collected
Number of previous DMT treatment | Baseline
  Number of previous DMT treatment will be collected
Line of previous DMT treatment | Baseline
  Line of previous DMT treatment will be collected
Type of previous DMT | Baseline
  Type of previous DMT will be collected:
  * Any interferon beta
  * Glatiramer acetate
  * Dimethyl fumarate
  * Teriflunomide
  * Fingolimod
  * Natalizumab
  * Cladribine
  * Alemtuzumab
  * Other B-cell therapy (Rituximab)
  * Other disease-modifying therapy
Percentage of participants with comorbidities | Baseline
  Percentage of participants with comorbidities will be collected:
  * Depression
  * Anxiety
  * Hypertension
  * Hypercholesterolemia
  * Chronic lung disease
  * Diabetes
  * Autoimmune disease
  * Migraine
  * Cancer (solid/blood)
  * Neurological Disease
  * Cardiovascular Disease
  * Other
Percentage of participants by number of comorbidities | Baseline
  Percentage of participants with 1, 2, 3 and more than 3 comorbidities will be collected
Percentage of smoking participants | Baseline
  Percentage of smoking participants will be collected
Percentage of alcohol intake participants | Baseline
  Percentage of alcohol intake participants will be collected
Percentage of patients by employment status | Baseline
  Percentage of patients by employment status (yes/no) will be collected
Percentage of participants by monthly income | Baseline
  Percentage of participants by monthly income (< 500$, 500-1000$, 1000-5000$, > 5000$) will be collected
Percentage of participants by educational level | Baseline
  Percentage of participants by educational level (college level, university level, none, other) will be collected
Percentage of participants by ethnicity | Baseline
  Percentage of participants by ethnicity will be collected:
  * Nationals
  * Non-Nationals, other Indian Bangladeshi Pakistani Egyptian Filipino Iranian Nepali Sri Lankan Chinese Other
Percentage of patients by frequency preference | Baseline
  Percentage of patients by frequency preference (daily, weekly, monthly, every 6 months, other) will be collected
Percentage of patients by route of administration | Baseline
  Percentage of patients by route of administration ( PO, IV, IM, SC) will be collected
Percentage of participants by type of coverage | Baseline
  Percentage of participants by type of coverage (Private, Governmental, Self-Payers, Others) will be collected

SECONDARY OUTCOMES:
Treatment Satisfaction Questionnaire for Medicines (TSQM) | baseline, 6 months, and 12 months
  TSQM, 1.4 Version (1.4) in English and Arabic will be used covering four areas of treatment-related satisfaction, which are safety, convenience, overall satisfaction, and effectiveness. The domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain
Total number of visits | 12 months
  Total number of visits will be collected
Number of visits to clinics | 12 months
  Number of visits to clinics will be collected
Reason for out patient department (OPD) visit | 12 months
  Reason for OPD visit will be collected
Number and reason of ER visits | 12 months
  Number and reason of Emergency Room (ER) visits will be collected
Number and reason of hospitalizations | 12 months
  Number and reason of hospitalizations will be collected
Length of hospital stay | 12 months
  Length of hospital stay (in days) will be collected
proxy costs for each visit | 12 months
  proxy costs for each visit by type and for all visits will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United Arab Emirates (5):
  - Novartis Investigative Site, Al Ain Abu Dhabi, United Arab Emirates
  - Novartis Investigative Site, Sharjah city, United Arab Emirates
  - Novartis Investigative Site, Abu Dhabi
  - Novartis Investigative Site, Dubai
  - Novartis Investigative Site, Sharjah city